CLINICAL TRIAL: NCT05051228
Title: Genetesis Accelerated Registry
Acronym: GEAR
Status: Suspended | Type: Observational
Why Stopped: Resourcing
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1000-05
Record Dates: First submitted 2021-01-28; First posted 2021-09-21 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Acute Myocardial Infarction; Acute Coronary Syndrome
Keywords: ischemia; acute myocardial injuries; CardioFlux; MCG; Cardiovascular disease
MeSH Terms: conditions — Acute Coronary Syndrome; Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- GEAR cohort: This is a noninvasive study that screens healthy and non-healthy volunteers for cardiovascular disease.
  Interventions: Device: CardioFlux

INTERVENTIONS:
Device: CardioFlux — Magnetocardiography (MCG) is a noninvasive method that measure the magnetic field that arises from the electrical activity of the heart cycle.

SUMMARY:
Heart disease is the number one cause of death in the United States, with over 650,000 deaths in 2019 alone. Many healthy individuals possess key risk factors for heart disease which include but are not limited to high blood pressure, high cholesterol, family history of heart disease, and diabetes. The purpose of the Genetesis Accelerated Registry (GEAR) study is to understand the potential for magnetocardiography to be utilized as a diagnostic, screening or surveillance tool for heart disease in healthy and non-healthy volunteers. Magnetocardiography (MCG) is a diagnostic method that analyzes and records the magnetic fields of the heart for the detection of various forms of heart disease. There will be a 12-month duration of the study where we propose to collect screening data from approximately 500 volunteers who present to the Genetesis facility for a 5-minute CardioFlux MCG scan. The volunteers will be contacted at intervals over a 1-year period for follow-up data and may choose whether or not they would like to provide follow-up data or participate in another scan.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of enrollment.

Exclusion Criteria:

1. < 18 years of age
2. Patients unable to fit into device
3. Non-ambulatory patients
4. Patients with present with or have reasonable clinical suspicion of any acute coronary syndrome for which delayed intervention could increase the risk or magnitude of damaged myocardium
5. Patients with claustrophobia or unable to lie supine for 5 minutes
6. Pregnant women
7. Poor candidate for follow-up (e.g. no access to phone)
8. Prisoners
9. Patients with a language barrier/language difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All volunteers presenting to the Genetesis facility (5950 Mason Montgomery Rd, Suite 1400, Mason, OH 45040) meeting the inclusion criteria for performance of a magnetocardiograph scan for diagnosis, risk assessment, or treatment monitoring due to cardiac illness (as determined by the Investigators) may participate. All other exclusion criteria are not specified contraindications for the device. If a patient has metal implants or implanted devices in your torso (e.g., pacemaker) or large amounts of implanted metal in other parts of their body, these may make their scan unreadable. There are no risks to the patient if they enter CardioFlux with metal. This scenario would simply require a re-scan, if the metal can be removed, or an unusable scan.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Cardioflux diagnosis/screening of ACS | 12 months
  Comparing the accuracy of Cardioflux to current standard of care when diagnosing/screening for ACS

CONTACTS AND LOCATIONS:
Locations (1):
- Genetesis Facility, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaikovsky I, Hailer B, Sosnytskyy V, Lutay M, Mjasnikov G, Kazmirchuk A, Bydnyk M, Lomakovskyy A, Sosnytskaja T. Predictive value of the complex magnetocardiographic index in patients with intermediate pretest probability of chronic coronary artery disease: results of a two-center study. Coron Artery Dis. 2014 Sep;25(6):474-84. doi: 10.1097/MCA.0000000000000107. PMID 24667125
- [Background] Hailer B, Chaikovsky I, Auth-Eisernitz S, Schafer H, Van Leeuwen P. The value of magnetocardiography in patients with and without relevant stenoses of the coronary arteries using an unshielded system. Pacing Clin Electrophysiol. 2005 Jan;28(1):8-16. doi: 10.1111/j.1540-8159.2005.09318.x. PMID 15660796
- [Background] Goernig M, Liehr M, Tute C, Schlosser M, Haueisen J, Figulla HR, Leder U. Magnetocardiography based spatiotemporal correlation analysis is superior to conventional ECG analysis for identifying myocardial injury. Ann Biomed Eng. 2009 Jan;37(1):107-11. doi: 10.1007/s10439-008-9598-5. Epub 2008 Nov 18. PMID 19015988
- [Background] Kwong JS, Leithauser B, Park JW, Yu CM. Diagnostic value of magnetocardiography in coronary artery disease and cardiac arrhythmias: a review of clinical data. Int J Cardiol. 2013 Sep 1;167(5):1835-42. doi: 10.1016/j.ijcard.2012.12.056. Epub 2013 Jan 19. PMID 23336954